CLINICAL TRIAL: NCT06351111
Title: Vagus Nerve Stimulation (VNS) in Spinal Cord Injury (SCI) Adaptive Follow-On Study
Acronym: SCI-AFOS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Dr. Seth Hays, Professor, The University of Texas at Dallas
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24-240; UG3NS131971 (NIH)
Record Dates: First submitted 2024-03-05; First posted 2024-04-08 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-04

CONDITIONS: SCI - Spinal Cord Injury
Keywords: SCI - Spinal Cord Injury; VNS - Vagus Nerve Stimulation; TPT - Targeted Plasticity Therapy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, open-label, adaptive, optional extension study model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Upper limb (UL) (Experimental): Participants in this arm will receive up to 36 sessions of VNS paired with upper limb rehabilitative exercises
  Interventions: Device: Active VNS
- Lower limb (LL) (Experimental): Participants in this arm will receive up to 36 sessions of VNS paired with lower limb rehabilitative exercises
  Interventions: Device: Active VNS
- Bladder control (BC) (Experimental): Participants in this arm will receive up to 36 sessions of VNS paired with bladder control rehabilitative exercises
  Interventions: Device: Active VNS
- Sensory (SY) (Experimental): Participants in this arm will receive up to 36 sessions of VNS paired with sensory rehabilitative exercises
  Interventions: Device: Active VNS

INTERVENTIONS:
Device: Active VNS — Subjects will receive active VNS paired with track-specific rehabilitation exercises.

SUMMARY:
This study is an open label extension of the SCI EFS clinical trial (NCT04288245) that developed an innovative strategy to enhance recovery of motor and sensory function after neurological injury. The objectives of this study are to provide continued safety assessment for the investigational ReStore system, and to gain further estimate of the effect of Vagus Nerve Stimulation (VNS) with rehabilitative exercises in four different tracks - upper limb (UL), lower limb (LL), bladder control (BC), and sensory (SY) for participants with chronic SCI (Spinal Cord Injury).

DETAILED DESCRIPTION:
A prospective, multi-center, non-randomized, open label extension of the SCI EFS trial (NCT04288245) participants implanted with the investigational ReStore Device for VNS Therapy. Following the completion of Phase 2 of the SCI EFS study, participants can enroll to one of the four tracks. Under each track, participants will undergo up to 36 sessions of rehabilitative exercises self-paced by participants with targeted completion of 3 sessions per week. Evaluations will be administered at the beginning and end of each track (additional progress checks may be conducted, as required by the staff) to monitor participant progress. Upon completion of a track, participants can choose to re-enroll in the same or a different track. Adverse events will be documented and assessed throughout the trial.

ELIGIBILITY:
General Inclusion Criteria:

1. Completed phase 2 of the SCI EFS study (NCT04288245)
2. Willing to comply with procedures for the entire duration of the study (study protocol compliance)
3. Provision of signed and dated informed consent form
4. Access to reliable communication and internet connections (for those intending to complete sessions at home)
5. Has not had their VNS device explanted

General Exclusion Criteria:

1. Concurrent participation in another active interventional trial or participation in an active interventional trial within 7 days prior to enrollment
2. Any medical condition or other circumstances that might interfere with their ability to return for follow-up visits in the judgment of the Investigator
3. Any condition which would preclude adequate evaluation of device's safety and performance in the judgment of the Investigator
4. Individuals who have a change in medical condition or health status such that they would meet the exclusion criteria of the EFS
5. Concomitant clinically significant brain injuries
6. Receiving any other therapy that would interfere with VNS
7. Females of childbearing potential who are either pregnant, lactating, heterosexually active, or planning to become pregnant or heterosexually active during study participation; and who are not using, or will not agree to use medically acceptable birth control methods
8. Psychiatric disorders, psychosocial, and/or cognitive impairment that would interfere with study participation, as assessed by medical evaluation
9. Participants with a current or past: (i) medical (psychiatric, non-psychiatric) condition, disease, disorder, injury, or disability; or (ii) non-medical situation or circumstance that, in the opinion of the principal investigator, study participation:

   1. May pose a significant or undue risk to the person;
   2. Make it unlikely the person will complete all the study requirements per protocol; or
   3. May adversely impact the integrity of the data or the validity of the study results
10. Participants with active neoplastic disease.
11. Participants with significant local circulatory problems, (e.g. thrombophlebitis and lymphedema, and clinically-significant hypotension or bradycardia).
12. Participants with any medical condition or other circumstances that might interfere with their ability to return for follow-up visits in the judgment of the Investigator.
13. Any condition which, in the judgment of the Investigator, would preclude adequate evaluation of device's safety and performance.
14. Aphasia and other cognitive deficits may be present but participants will be excluded if are unable to understand the potential risks and benefits of the study or personally provide informed consent.
15. A recent history of syncope
16. A recent history of dysphagia
17. Currently require, or are likely to require diathermy
18. Significant respiratory issues that would interfere with participation
19. Non-English speaking
20. Patients who are acutely suicidal and/or have been admitted for a suicide attempt
21. As determined by the principal investigator, is under current incarceration or legal detention

Track Specific Inclusion Criteria:

Upper Limb (UL):

1)None

Lower Limb (LL):

1)Ambulatory with gait impairment

Bladder Control (BC):

1)Issues with urinary function arising from SCI, with partial voluntary initiation of voiding 2)Intermittent catheterization for bladder management

Sensory (SY):

1)Impairment in sensory function, based on the baseline assessments below:

1. US-NSA score <92 points
2. Two-point discrimination fingertip score >5mm
3. Two-point discrimination palm score >15mm
4. Tactile Discrimination Test score <16points
5. Semmes-Weinstein Monofilaments score >3.61g

   Track Specific Exclusion Criteria:

   Upper Limb (UL):

   1)None

   Lower Limb (LL):

   1)None

   Bladder Control (BC):

   1)Indwelling catheter use 2)Participants with a history of severe or recurrent autonomic dysreflexia 3)Technical limitations that would preclude bladder ultrasonography assessments 4)Medical history that would preclude adequate evaluation of urologic outcomes

   Sensory (SY):
   1. Pain that would impede study participation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (device safety) | Starting at session 1 on week 1, throughout the study up to last session 36 on week 15.
  UL, LL, BC and SY - Review of adverse events reported throughout the trial will be used to inform the potential risks associated with the ReStore System

SECONDARY OUTCOMES:
Jebsen-Taylor Hand Function (JTHF) Score | At session 1 on week 1, session 36 on week 15, and as needed during intervening sessions from week 2 to 14.
  UL only - Determine whether VNS therapy improves Jebsen-Taylor Hand Function (JTHF) score compared to baseline. This measure is not a scale. Each item is timed from 0 to 120 seconds. Lower/faster values are better.
Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) | At session 1 on week 1, session 36 on week 15, and as needed during intervening sessions from week 2 to 14.
  UL only - Determine whether VNS therapy improves the GRASSP score compared to baseline. This scale is from 0 to 116 points. Higher scores are better.
Force & Range of motion | At session 1 on week 1, session 36 on week 15, and as needed during intervening sessions from week 2 to 14.
  UL only - Determine whether VNS therapy improves force and range of motion in the hand and wrist compared to baseline.
6 Meter Walk Test (6MWT) | At session 1 on week 1, session 36 on week 15, and as needed during intervening sessions from week 2 to 14.
  LL only - Determine whether VNS therapy improves six-minute walking test (6MWT) score compared to baseline. This measure is not a scale. Higher distance covered is better.
10 Meter Walk Test (10MWT) | At session 1 on week 1, session 36 on week 15, and as needed during intervening sessions from week 2 to 14.
  LL only - Determine whether VNS therapy improves 10-Meter Walk Test (10-MWT) score compared to baseline. This measure is not a scale. Lower time to complete is better.
Walking Index for Spinal Cord Injury II (WISCI II) | At session 1 on week 1, session 36 on week 15, and as needed during intervening sessions from week 2 to 14.
  LL only - Determine whether VNS therapy improves Walking Index for Spinal Cord Injury II (WISCI II) score compared to baseline. This scale is from 0-20. Higher scores are better.
Berg's Balance Scale (BBG) | At session 1 on week 1, session 36 on week 15, and as needed during intervening sessions from week 2 to 14.
  LL only - Determine whether VNS therapy improves Berg's Balance Scale (BBG) score compared to baseline. This scale is from 0 to 56. Higher scores are better.
Timed Up-and Go (TUG)Test | At session 1 on week 1, session 36 on week 15, and as needed during intervening sessions from week 2 to 14.
  LL only - Determine whether VNS therapy improves Timed Up-and Go (TUG)Test score compared to baseline. This measure is not a scale. Lower time to complete is better.
Lower Extremity Motor Score (LEMS) | At session 1 on week 1, session 36 on week 15, and as needed during intervening sessions from week 2 to 14.
  LL only - Determine whether VNS therapy improves Lower Extremity Motor Score (LEMS) compared to baseline. This scale is from 0 to 50. Higher scores are better.
Voiding efficiency | At session 1 on week 1, session 36 on week 13, and as needed during intervening sessions on week 2 to 13.
  BC only - Estimate the shift in voiding efficiency through bladder ultrasonography assessment following active VNS
Bladder volume capacity | At session 1 on week 1, session 36 on week 13, and as needed during intervening sessions on week 2 to 13.
  BC only - Estimate the shift in bladder volume capacity during bladder ultrasonography assessment following active VNS
Postvoid residual volume (PVR) | At session 1 on week 1, session 36 on week 13, and as needed during intervening sessions on week 2 to 13.
  BC only - Estimate the shift in PVR during bladder ultrasonography assessment following active VNS
Neurogenic Bladder Symptom Score (NBSS) questionnaire | At session 1 on week 1, session 36 on week 13, and as needed during intervening sessions on week 2 to 13.
  BC only - Estimate the shift in NBSS score following active VNS. This scale is from 0 to 78. Lower scores are better.
Urinary Distress Inventory (UDI-6), short form questionnaire | At session 1 on week 1, session 36 on week 13, and as needed during intervening sessions on week 2 to 13.
  BC only - Estimate the shift in the UDI-6 questionnaire score following active VNS. This scale is from 0 to 18. Lower scores are better.
Two - Point Discrimination | At session 1 on week 1, on week 8, week 12 and as needed during intervening sessions from week 2 to 7.
  SY only - Determine whether VNS therapy improves Two-Point Discrimination (2PD) score compared to baseline. This measure is not a scale but the ability to feel two separate points of touch on the skin instead of just one. It's a sensory test used in neurological exams to assess the density and health of nerve innervation in a specific area of the body. The test involves determining the smallest distance between two points that a person can still perceive as two separate stimuli.
Tactile Discrimination Test (TDT) | At session 1 on week 1, on week 8, week 12, and as needed during intervening sessions from week 2 to 7.
  SY only- Determine whether VNS therapy improves Tactile Discrimination Test (TDT) score compared to baseline. This scale is from 0 to 25 points. Higher scores are better.
Semmes-Weinstein Monofilaments (SWM) | At session 1 on week 1, on week 8, week 12, and as needed during intervening sessions from week 2 to 7.
  SY only - Determine whether VNS therapy improves Semmes-Weinstein Monofilaments (SWM) test score compared to baseline. This measure is not a scale but a test to assess a person's light touch sensation using a set of filaments of different thickness to identify loss of protective sensation in areas like feet or hands. The level of the filament required to elicit a response provides a measurement of the patient's sensory threshold. Thinner filament indicates better sensory function.
US-Nottingham Sensory Assessment (US-NSA) | At session 1 on week 1, on week 8, week 12, and as needed during intervening sessions from week 2 to 7.
  SY only - Determine whether VNS therapy improves US-Nottingham Sensory Assessment (US-NSA) score compared to baseline. This assessment is a scale ranging from 0 to 92 for the upper extremity, and 0 to 172 for the combined upper and lower extremities. Higher scores indicate better sensory function.
International SCI Pain Basic Data | At session 1 on week 1, on week 8, week 12, and as needed during intervening sessions from week 2 to 7.
  SY only- Determine whether VNS therapy can reduce pain severity and improve patient-reported outcomes of the International SCI Pain Basic Data Set, compared to baseline measures. This measure uses a numeric rating scale from 0 to 10, where 0 indicates no pain. Lower scores indicate lower pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Wigginton, Principal Investigator — The University of Texas at Dallas; Robert Rennaker, Principal Investigator — The University of Texas at Dallas; Rita Hamilton, Principal Investigator — Baylor Scott and White Institute for Rehabilitation
Locations (2):
- United States (2):
  - Baylor University Medical Center, Dallas, Texas
  - Texas Biomedical Device Center, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No